CLINICAL TRIAL: NCT01839656
Title: A Study to Assess the Efficacy, Safety, Tolerability, and Pharmacokinetics of Multiple Doses of ISIS 396443 Delivered Intrathecally to Patients With Infantile-Onset Spinal Muscular Atrophy
Brief Title: A Study to Assess the Efficacy, Safety and Pharmacokinetics of Nusinersen (ISIS 396443) in Infants With Spinal Muscular Atrophy (SMA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 396443-CS3A; 2017-000621-12 (EudraCT Number)
Expanded Access: NCT02865109 (No longer available)
Record Dates: First submitted 2013-04-22; First posted 2013-04-25 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; SMA; SMN; SMNRx; ISIS-SMNRx; ISIS 396443; IONIS-SMNRx; Spinraza; Nusinersen
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nusinersen 6 mg (Experimental)
  Interventions: Drug: nusinersen
- Nusinersen 12 mg (Experimental)
  Interventions: Drug: nusinersen

INTERVENTIONS:
Drug: nusinersen — Administered by intrathecal (IT) injection
  Other Names: ISIS 396443; Spinraza; BIIB058; IONIS SMN Rx; ISIS SMNRx

SUMMARY:
The primary objective is to examine the clinical efficacy of multiple doses of nusinersen (ISIS 396443) administered intrathecally to participants with Infantile-Onset Spinal Muscular Atrophy (SMA). The secondary objectives are to examine the safety and tolerability of multiple doses of nusinersen administered intrathecally to participants with infantile-onset SMA and to examine the cerebral spinal fluid (CSF) and plasma Pharmacokinetics (PK) of multiple doses of nusinersen administered intrathecally to participants with infantile-onset SMA.

DETAILED DESCRIPTION:
This study was conducted and the protocol was registered by Ionis Pharmaceuticals, Inc.. In August 2016, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Genetic documentation of 5q SMA (homozygous gene deletion or mutation)
* Onset of clinical signs and symptoms consistent with SMA at ≥ 21 days and <6 months (180 days) of age
* At study entry, receiving adequate nutrition and hydration (with or without gastrostomy), in the opinion of the Site Investigator
* Body weight >5th percentile for age using Center of Disease Control and Prevention (CDC) guidelines
* Medical care meets and is expected to continue to meet guidelines set out in the Consensus Statement for Standard of Care in SMA (Wang et al. 2007), in the opinion of the Site Investigator
* Gestational age of 35 to 42 weeks and gestation body weight ≥2 kg
* Reside within approximately 9 hours ground-travel distance from a participating study center for the duration of the study. Residence >2 hours ground-travel distance from a study center must obtain clearance from the Site Investigator and the study Medical Monitor
* Able to complete all study procedures, measurements and visits and parent or guardian/participant has adequately supportive psychosocial circumstances, in the opinion of the Site Investigator

Exclusion Criteria:

* Hypoxemia (O2 saturation awake <96% or O2 saturation asleep <96%, without ventilation support)
* Presence of an untreated or inadequately treated active infection requiring systemic antiviral or antimicrobial therapy at any time during the screening period
* History of brain or spinal cord disease that would interfere with the lumbar puncture (LP) procedures, CSF circulation, or safety assessments
* Presence of an implanted shunt for the drainage of cerebrospinal fluid (CSF) or an implanted central nervous system (CNS) catheter
* History of bacterial meningitis
* Clinically significant abnormalities in hematology or clinical chemistry parameters, as assessed by the Site Investigator, at screening that would render the participant unsuitable for inclusion
* Treatment with another investigational drug (e.g., albuterol, riluzole, carnitine, creatine, sodium phenylbutyrate, salbutamol, valproate, hydroxyurea etc), biological agent, or device within 90 days prior to enrollment or anytime during the study. Any history of gene therapy or cell transplantation
* The participants parent(s) or legal guardian(s) is unable to understand the nature, scope, and possible consequences of the study, or does not agree to comply with the protocol defined schedule of assessments
* Ongoing medical condition that according to the Site Investigator would interfere with the conduct and assessments of the study. Examples are medical disability other than SMA that would interfere with the assessment of safety or would compromise the ability of the participant to undergo study procedures

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 21 Days to 210 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2013-05-08 (Actual); Primary Completion 2017-08-21 (Actual); Study Completion 2017-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (4):
- United States (3):
  - Stanford University Medical Center, Stanford, California
  - Nemours Children's Hospital, Orlando, Florida
  - Columbia University Medical Center, New York, New York
- The Hospital for Sick Children (SickKids), Toronto, Ontario, Canada

REFERENCES:
- [Derived] Finkel RS, Chiriboga CA, Vajsar J, Day JW, Montes J, De Vivo DC, Bishop KM, Foster R, Liu Y, Ramirez-Schrempp D, Schneider E, Bennett CF, Wong J, Farwell W. Treatment of infantile-onset spinal muscular atrophy with nusinersen: final report of a phase 2, open-label, multicentre, dose-escalation study. Lancet Child Adolesc Health. 2021 Jul;5(7):491-500. doi: 10.1016/S2352-4642(21)00100-0. Epub 2021 Jun 3. PMID 34089650
- [Derived] Darras BT, Farrar MA, Mercuri E, Finkel RS, Foster R, Hughes SG, Bhan I, Farwell W, Gheuens S. An Integrated Safety Analysis of Infants and Children with Symptomatic Spinal Muscular Atrophy (SMA) Treated with Nusinersen in Seven Clinical Trials. CNS Drugs. 2019 Sep;33(9):919-932. doi: 10.1007/s40263-019-00656-w. PMID 31420846
- [Derived] Finkel RS, Chiriboga CA, Vajsar J, Day JW, Montes J, De Vivo DC, Yamashita M, Rigo F, Hung G, Schneider E, Norris DA, Xia S, Bennett CF, Bishop KM. Treatment of infantile-onset spinal muscular atrophy with nusinersen: a phase 2, open-label, dose-escalation study. Lancet. 2016 Dec 17;388(10063):3017-3026. doi: 10.1016/S0140-6736(16)31408-8. Epub 2016 Dec 7. PMID 27939059
- See also: Cure SMA — http://www.curesma.org
- See also: Muscular Dystrophy Association — http://mda.org/disease/spinal-muscular-atrophy
- See also: National Organization for Rare Diseases — https://www.rarediseases.org
- See also: Clinical Study Report (CSR) Synopsis - a results summary — http://clinicalresearch.biogen.com/Content/Studies/CS3A_Biogen.com%20Packet_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 23 participants screened, 2 were screening failures. A total of 21 participants enrolled; 1 was withdrawn from the study due to respiratory failure prior to receiving the first dose of study treatment. Twenty participants received at least 1 dose of study treatment and were included in the efficacy, safety, and PK analyses.
Groups:
- Nusinersen 6 mg: Participants received nusinersen 6 mg injections as an intrathecal (IT) bolus through a lumbar puncture (LP) on Days 1, 15, and 85. Maintenance doses of 12 mg were given on Days 253, 379, 505, 631, 757, 883, 1009, 1135, and 1261.
- Nusinersen 12 mg: Participants received nusinersen 12 mg injections as an intrathecal (IT) bolus through a lumbar puncture (LP) on Days 1, 15, and 85. Maintenance doses of 12 mg were given on Days 253, 379, 505, 631, 757, 883, 1009, 1135, and 1261.
Period: Overall Study
Arm/Group | Nusinersen 6 mg | Nusinersen 12 mg
Started | 5 | 16
Completed Loading Dose Period | 4 | 15
Completed | 2 | 0
Not Completed | 3 | 16
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse event, serious fatal | 1 | 4
Not completed — Early study closure | 0 | 11
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nusinersen 6 mg | Nusinersen 12 mg | Total
Number analyzed (Participants) | 4 | 16 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 16 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 8
  Male | 3 | 9 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 15 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 13 | 16
  Black | 0 | 1 | 1
  Asian | 0 | 1 | 1
  American Indian or Alaskan Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Multiple Race | 1 | 0 | 1
  Other | 0 | 1 | 1
Hammersmith Infant Neurological Examination (HINE) Head Control Motor Milestones at Baseline [Count of Participants; unit: Participants] — Baseline was defined as the last non-missing value prior to the first dose of nusinersen.
  Participants
    Unable to maintain head upright | 3 | 13 | 16
    Wobbles | 1 | 2 | 3
    All the time maintained upright | 0 | 1 | 1
HINE Sitting Motor Milestones at Baseline [Count of Participants; unit: Participants] — Baseline was defined as the last non-missing value prior to the first dose of nusinersen.
  Participants
    Cannot sit | 4 | 15 | 19
    Sits with support at hips | 0 | 1 | 1
    Props | 0 | 0 | 0
    Stable sit | 0 | 0 | 0
    Pivots (rotates) | 0 | 0 | 0
HINE Voluntary Grasp Motor Milestones at Baseline [Count of Participants; unit: Participants] — Baseline was defined as the last non-missing value prior to the first dose of nusinersen.
  Participants
    No grasp | 0 | 3 | 3
    Uses whole hand | 4 | 13 | 17
    Index finger and thumb but immature grasp | 0 | 0 | 0
    Pincer grasp | 0 | 0 | 0
HINE Ability to Kick Motor Milestones at Baseline [Count of Participants; unit: Participants] — Baseline was defined as the last non-missing value prior to the first dose of nusinersen.
  Participants
    No kicking | 1 | 5 | 6
    Kick horizontally, legs do not lift | 3 | 10 | 13
    Upward (vertically) | 0 | 1 | 1
    Touches leg | 0 | 0 | 0
    Touches toes | 0 | 0 | 0
HINE Rolling Motor Milestones at Baseline [Count of Participants; unit: Participants] — Baseline was defined as the last non-missing value prior to the first dose of nusinersen.
  Participants
    No rolling | 4 | 15 | 19
    Rolling side to side | 0 | 0 | 0
    Prone to supine | 0 | 1 | 1
    Supine to prone | 0 | 0 | 0
HINE Crawling Motor Milestones at Baseline [Count of Participants; unit: Participants] — Baseline was defined as the last non-missing value prior to the first dose of nusinersen.
  Participants
    Does not lift head | 4 | 14 | 18
    On elbow | 0 | 1 | 1
    On outstretched hand | 0 | 1 | 1
    Crawling flat on abdomen | 0 | 0 | 0
    Crawling on hands and knees | 0 | 0 | 0
HINE Standing Motor Milestones at Baseline [Count of Participants; unit: Participants] — Baseline was defined as the last non-missing value prior to the first dose of nusinersen.
  Participants
    Does not support weight | 4 | 15 | 19
    Supports weight | 0 | 1 | 1
    Stands with support | 0 | 0 | 0
    Stands unaided | 0 | 0 | 0
HINE Walking Motor Milestones at Baseline [Count of Participants; unit: Participants] — Baseline was defined as the last non-missing value prior to the first dose of nusinersen.
  Participants
    No walking | 4 | 15 | 19
    Bouncing | 0 | 1 | 1
    Cruising (walks holding on) | 0 | 0 | 0
    Walking independently | 0 | 0 | 0
Distribution of Total Scores of the CHOP-INTEND Scale at Baseline [Count of Participants; unit: Participants] — The Children's Hospital of Philadelphia Infant Test for Neuromuscular Disease (CHOP-INTEND) test includes 16 items structured to move from easiest to hardest with the grading including gravity eliminated (lower scores) to antigravity movements (higher scores). All item scores range from 0 (worst) to 4 (best). Total scores range from 0 to 64, with higher scores indicating better movement functioning. Baseline was defined as the last non-missing value prior to the first dose of nusinersen.
  Participants
    0 to 9 | 0 | 0 | 0
    10 to 19 | 0 | 2 | 2
    20 to 29 | 3 | 6 | 9
    30 to 39 | 1 | 6 | 7
    40 to 49 | 0 | 1 | 1
    50 to 59 | 0 | 0 | 0
    60 to 64 | 0 | 1 | 1
Mean CHOP INTEND Total Scores at Baseline [Mean (Standard Deviation); unit: Units on a scale] — The CHOP-INTEND test includes 16 items structured to move from easiest to hardest with the grading including gravity eliminated (lower scores) to antigravity movements (higher scores). All item scores range from 0 (worst) to 4 (best). Total scores range from 0 to 64, with higher scores indicating better movement functioning. Baseline was defined as the last non-missing value prior to the first dose of nusinersen.
  Units on a scale | 27 (5) | 30 (12) | 30 (11)
Mean Compound Muscle Action Potential (CMAP) Amplitude of the Peroneal Nerve at Baseline [Mean (Standard Deviation); unit: millivolts (mV)] — Baseline was defined as the last non-missing value prior to the first dose of nusinersen.
  millivolts (mV) | 0.673 (0.501) | 0.518 (0.664) | 0.549 (0.626)
Mean CMAP Amplitude of the Ulnar Nerve at Baseline [Mean (Standard Deviation); unit: mV] — Baseline was defined as the last non-missing value prior to the first dose of nusinersen.
  mV | 0.372 (0.177) | 0.532 (0.878) | 0.501 (0.786)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Achieved Improvement in Motor Milestones as Assessed by Section 2 of the HINE at the Last Visit
Description: Section 2 of HINE consists of 8 independent milestone categories. Within each of these categories, participants can progress from complete absence of a motor ability (the lowest level in each category) through multiple milestones (2 to 4 levels in each category) to the highest level within the category. Overall, there are a total of 26 milestones that can be achieved across the 8 categories. Improvement was defined as any of the following: 1. An increase from baseline of 2 milestones or more, or the achievement of pincer grasp in the voluntary grasp category 2. An increase from baseline of 2 milestones or more, or achievement of touching toes in the ability to kick category 3. An increase from baseline of 1 milestone or more in any of the remaining 6 categories: head control, rolling, sitting, crawling, standing, or walking.
Time Frame: Day 1352 or Early Termination
Population: Safety Population: All participants who were registered and received at least 1 dose of nusinersen.
Measure: Number; unit: Percent of participants
Arm/Group | Nusinersen 6 mg | Nusinersen 12 mg
Number analyzed (Participants) | 4 | 16
Percent of participants | 25.0 | 68.8

2. Secondary Outcome: Event-free Survival at the End of Study
Description: Event-free survival was defined as the percent of participants who were alive and did not require permanent ventilatory support (defined as tracheostomy or the need for ≥16 hours ventilation/day continuously for at least 2 weeks in the absence of an acute reversible illness) Event-free survival was estimated using Kaplan-Meier methodology.
Time Frame: Up to Day 1638
Population: Safety Population: All participants who were registered and received at least 1 dose of nusinersen.
Measure: Number; unit: Percent of participants
Arm/Group | Nusinersen 6 mg | Nusinersen 12 mg
Number analyzed (Participants) | 4 | 16
Percent of participants | 25.0 | 62.5

3. Secondary Outcome: Percent of Participants With Improved Motor Function at the Last Visit as Assessed by the CHOP-INTEND Motor Function Scale
Description: The CHOP-INTEND test includes 16 items structured to move from easiest to hardest with the grading including gravity eliminated (lower scores) to antigravity movements (higher scores). All item scores range from 0 (worst) to 4 (best). Total scores range from 0 to 64, with higher scores indicating better movement functioning. Improvement was defined as an increase in total CHOP INTEND score ≥4 points from baseline as of the last study visit.
Time Frame: Day 1352 or Early Termination
Population: Safety Population: All participants who were registered and received at least 1 dose of nusinersen.
Measure: Number; unit: Percent of participants
Arm/Group | Nusinersen 6 mg | Nusinersen 12 mg
Number analyzed (Participants) | 4 | 16
Percent of participants | 25.0 | 62.5

4. Secondary Outcome: Change in Neuromuscular Electrophysiology at the Last Visit as Assessed by the Change From Baseline in CMAP Amplitude
Description: CMAP is an electrophysiological technique that can be used to determine the approximate number of motor neurons in a muscle or group of muscles. A positive change from Baseline indicates that the number of motor neurons increased.
Time Frame: Baseline, Day 1072
Population: Safety Population: All participants who were registered and received at least 1 dose of nusinersen. Here, number of participants analyzed is the participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Nusinersen 6 mg | Nusinersen 12 mg
Number analyzed (Participants) | 2 | 8
mV
  Peroneal nerve | 1.88 (2.58) | 2.81 (1.28)
  Ulnar nerve | 0.776 (1.448) | 0.685 (0.415)

5. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs) and/or Serious Adverse Events (SAEs)
Description: AE: any unfavorable and unintended sign, symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product. SAE: any AE that in the view of either the Investigator or Sponsor, meets any of the following criteria: results in death; is life threatening: that is, poses an immediate risk of death at the time of the event; requires in-patient hospitalization or prolongation of existing hospitalization; results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; results in congenital anomaly or birth defect in the offspring of the subject (whether male or female); is an important medical event in the opinion of the Investigator or Sponsor.
Time Frame: Up to Day 1352
Population: Safety Population: All participants who were registered and received at least 1 dose of nusinersen.
Measure: Number; unit: participants
Arm/Group | Nusinersen 6 mg | Nusinersen 12 mg
Number analyzed (Participants) | 4 | 16
participants
  Any AE | 4 | 16
  Any SAE | 3 | 13

6. Secondary Outcome: Concentration of Nusinersen in Cerebrospinal Fluid (CSF)
Description: The concentration of nusinersen in CSF was measured by using standard laboratory assays.
Time Frame: Day 1135 (Predose)
Population: PK Population: All participants who were registered and had at least 1 evaluable postdose PK sample. Here, number of participants analyzed is the participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Nusinersen 6 mg | Nusinersen 12 mg
Number analyzed (Participants) | 2 | 6
nanograms/milliliter (ng/mL) | 12.2 (8.60) | 11.1 (4.99)

7. Secondary Outcome: PK Parameters of Nusinersen in Plasma: Maximum Concentration (Cmax)
Description: Cmax is the maximum observed concentration of study drug in plasma.
Time Frame: Day 1 (Predose and 1, 2, and 4 hours [hr] Postdose) and Day 2 (24 hr Postdose )
Population: PK Population: All participants who were registered and had at least 1 evaluable postdose PK sample.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nusinersen 6 mg | Nusinersen 12 mg
Number analyzed (Participants) | 4 | 16
ng/mL | 396 (311) | 829 (625)

8. Secondary Outcome: PK Parameters of Nusinersen in Plasma: Time to Reach Cmax (Tmax)
Description: Tmax is the time at which Cmax occurs.
Time Frame: Day 1 (Predose and 1, 2, and 4 hours [hr] Postdose) and Day 2 (24 hr Postdose )
Population: PK Population: All participants who were registered and had at least 1 evaluable postdose PK sample.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Nusinersen 6 mg | Nusinersen 12 mg
Number analyzed (Participants) | 4 | 16
hr | 2.09 (1.35) | 2.37 (1.25)

9. Secondary Outcome: PK Parameters of Nusinersen in Plasma: Area Under the Plasma Concentrations Time Curve From the Time of the IT Dose to Four Hours After Dosing (AUC0-4)
Description: AUC is area under the plasma concentration-time curve from zero time (Predose) to 4 hours after IT administration of study drug. AUC was determined by using the linear trapezoidal rule.
Time Frame: Day 1 (Predose and 1, 2, and 4 hours [hr] Postdose) and Day 2 (24 hr Postdose )
Population: PK Population: All participants who were registered and had at least 1 evaluable postdose PK sample.
Measure: Mean (Standard Deviation); unit: ng x hr/mL
Arm/Group | Nusinersen 6 mg | Nusinersen 12 mg
Number analyzed (Participants) | 4 | 16
ng x hr/mL | 894 (610) | 2181 (1488)

ADVERSE EVENTS:
Time Frame: Up to Day 1359
Groups:
- Nusinersen 12 mg: Participants aged 21 days to 7 months old with infantile-onset SMA received nusinersen 12 mg injections at regular intervals for up to 45 months.
Arm/Group | Nusinersen 6 mg | Nusinersen 12 mg
All-Cause Mortality (participants affected / at risk) | 1/4 | 4/16
Serious Adverse Events (participants affected / at risk) | 3/4 | 13/16
Other Adverse Events (participants affected / at risk) | 4/4 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nusinersen 6 mg (N=4) | Nusinersen 12 mg (N=16)
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 1
Pneumopericardium (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Adenovirus infection (Infections and infestations) | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 3
Corona virus infection (Infections and infestations) | 1 | 1
Enterovirus infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1
Metapneumovirus infection (Infections and infestations) | 0 | 2
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 5
Pneumonia adenoviral (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 1
Pneumonia pseudomonas aeruginosa (Infections and infestations) | 1 | 1
Pneumonia viral (Infections and infestations) | 0 | 3
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 3
Respiratory tract infection (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nusinersen 6 mg (N=4) | Nusinersen 12 mg (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 2
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Clinodactyly (Congenital, familial and genetic disorders) | 0 | 1
Cryptorchism (Congenital, familial and genetic disorders) | 1 | 1
High arched palate (Congenital, familial and genetic disorders) | 1 | 0
Hip dysplasia (Congenital, familial and genetic disorders) | 0 | 1
Pectus carinatum (Congenital, familial and genetic disorders) | 0 | 1
Plagiocephaly (Congenital, familial and genetic disorders) | 1 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 1
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1
Astigmatism (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Erythema of eyelid (Eye disorders) | 0 | 1
Eye irritation (Eye disorders) | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 8
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Flatulence (Gastrointestinal disorders) | 1 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 6
Haematemesis (Gastrointestinal disorders) | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 1
Teething (Gastrointestinal disorders) | 2 | 2
Tongue atrophy (Gastrointestinal disorders) | 0 | 2
Tooth crowding (Gastrointestinal disorders) | 1 | 0
Traumatic tooth displacement (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 5
Cyst (General disorders) | 0 | 1
Device leakage (General disorders) | 0 | 1
Device occlusion (General disorders) | 0 | 1
Discomfort (General disorders) | 1 | 1
Infusion site extravasation (General disorders) | 0 | 1
Injection site bruising (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 2 | 3
Pain (General disorders) | 0 | 4
Pyrexia (General disorders) | 3 | 14
Vessel puncture site bruise (General disorders) | 0 | 1
Vessel puncture site haemorrhage (General disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 3
Adenoviral upper respiratory infection (Infections and infestations) | 0 | 1
Adenovirus infection (Infections and infestations) | 0 | 1
Bacterial disease carrier (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Bacterial tracheitis (Infections and infestations) | 0 | 2
Bronchiolitis (Infections and infestations) | 0 | 1
Candida nappy rash (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 0 | 3
Enterovirus infection (Infections and infestations) | 0 | 2
Erythema infectiosum (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 1
Gastritis viral (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Haemophilus infection (Infections and infestations) | 0 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Moraxella infection (Infections and infestations) | 0 | 1
Mucocutaneous candidiasis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 7
Oral candidiasis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 6
Parainfluenzae virus infection (Infections and infestations) | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 5
Pneumonia moraxella (Infections and infestations) | 0 | 1
Pneumonia pseudomonas aeruginosa (Infections and infestations) | 1 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 3 | 4
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 3
Rhinovirus infection (Infections and infestations) | 0 | 4
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 10
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 4
Viral rash (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Ear abrasion (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 2
Feeding tube complication (Injury, poisoning and procedural complications) | 0 | 3
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 3
Laceration (Injury, poisoning and procedural complications) | 0 | 2
Lip injury (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Post gastric surgery syndrome (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Tooth injury (Injury, poisoning and procedural complications) | 0 | 1
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 | 0
Bacterial test positive (Investigations) | 1 | 0
Bone density decreased (Investigations) | 0 | 2
Breath sounds abnormal (Investigations) | 0 | 1
Heart rate decreased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 0 | 1
Human rhinovirus test positive (Investigations) | 0 | 3
Moraxella test positive (Investigations) | 0 | 1
Neutrophil count increased (Investigations) | 0 | 2
Neutrophil percentage increased (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 2
Pseudomonas test positive (Investigations) | 0 | 1
Serratia test positive (Investigations) | 0 | 1
Staphylococcus test positive (Investigations) | 0 | 1
Streptococcus test positive (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 1
White blood cell count increased (Investigations) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Hypophagia (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 1
Weight gain poor (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Deformity thorax (Musculoskeletal and connective tissue disorders) | 1 | 2
Hand deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 3 | 7
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Kyphoscoliosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Kyphosis (Musculoskeletal and connective tissue disorders) | 2 | 3
Lordosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Rib deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 2 | 6
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 2 | 2
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Drooling (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hyporeflexia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Muscle contractions involuntary (Nervous system disorders) | 1 | 3
Nystagmus (Nervous system disorders) | 1 | 0
Speech disorder developmental (Nervous system disorders) | 1 | 2
Syncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 3
Expressive language disorder (Psychiatric disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Laryngeal granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tracheal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 3
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 | 3
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 5
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1
Capillary fragility (Vascular disorders) | 0 | 1
Essential hypertension (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Subgaleal haematoma (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2016-01-25): https://cdn.clinicaltrials.gov/large-docs/56/NCT01839656/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT01839656/SAP_001.pdf